CLINICAL TRIAL: NCT06606106
Title: A Multiple-Ascending Dose Study to Investigate the Safety, Pharmacokinetics, and Pharmacodynamics of LY3537031 in Overweight and Obese Participants and Healthy Volunteers
Brief Title: A Study of LY3537031 in Overweight, Obese, and Healthy Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 27199; J2S-MC-GZMD (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-08-27; First posted 2024-09-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- LY3537031 Part A (Cohorts 1-7) (Experimental): Multiple-ascending doses of LY3537031 administered subcutaneously (SC)
  Interventions: Drug: LY3537031
- Placebo Part A (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo
- LY3537031 Part B (Cohorts 8-11) (Experimental): Multiple-ascending doses of LY3537031 administered SC
  Interventions: Drug: LY3537031
- Placebo Part B (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo
- LY3537031 Part C (Cohorts 12-15) (Experimental): Multiple-ascending doses of LY3537031 administered SC
  Interventions: Drug: LY3537031
- Placebo Part C (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo
- LY3537031 Part D (Cohorts 16-19) (Experimental): Multiple-ascending doses of LY3537031 administered SC
  Interventions: Drug: LY3537031
- Placebo Part D (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3537031 — Administered SC
  Arms: LY3537031 Part A (Cohorts 1-7); LY3537031 Part B (Cohorts 8-11); LY3537031 Part C (Cohorts 12-15); LY3537031 Part D (Cohorts 16-19)
Drug: Placebo — Administered SC
  Arms: Placebo Part A; Placebo Part B; Placebo Part C; Placebo Part D

SUMMARY:
This is a 4-part study that includes a Part A, Part B, Part C, and Part D. Parts A and D will study the safety and tolerability of the study drug known as LY3537031 in participants who are overweight and obese. Part B and Part C will study the safety and tolerability of LY3537031 in healthy participants. Part C will contain only Japanese and Chinese healthy participants.

Blood tests will be performed to check how much LY3537031 gets into the bloodstream and how long it takes the body to eliminate it. Body weight will be measured. The study will last approximately 49 weeks excluding a screening period.

ELIGIBILITY:
Inclusion Criteria:

* Have a BMI within the range of:

  * Parts A and D: 27.0 to 45.0 kilogram per square meter (kg/m²)
  * Parts B and C: 22.0 to 26.9 kg/m²
* Parts B and C: Weigh 60 kg (80 pounds (lbs)) or more at screening
* Have no significant (not more than 5%) self-reported weight gain or loss in the past 3 months prior to screening
* Have a thyroid stimulating hormone (TSH) value within normal local laboratory ranges.

Exclusion Criteria:

* Have undergone any form of bariatric surgery
* Participants who are lactating
* Have taken medications that promote weight loss within 90 days before screening
* Have a serum calcitonin level (at screening) of greater than or equal to 35 nanograms per liter (ng/L) (35 picograms per milliliter (pg/mL), 10.2 picomoles per liter (pmol/L))

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs), Serious Adverse Event(s) (SAEs), and Adverse Event(s) (AEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline to Study Completion (Up to 56 Weeks)
  A summary of TEAEs, SAEs, and AEs regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3537031 | Predose on Day 1 through Week 56
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3537031 | Predose on Day 1 through Week 56
Pharmacodynamic (PD): Change from Baseline in Body Weight | Baseline up to Week 56
PD: Change from Baseline in Fasting Glucose | Baseline up to Week 56
PD: Change from Baseline in Oral Glucose Tolerance Test (OGTT) Results | Baseline up to Week 56
PD: Change from Baseline in AUC of Glucose | Baseline Up to Week 56
PD: Change from Baseline in Insulin Levels | Baseline Up to Week 56
PD: Change from Baseline in Connecting Peptide (C-peptide) Levels | Baseline Up to Week 56
PD: Change from Baseline in Cmax of Acetaminophen to Assess the Delay in Gastric Emptying | Baseline up to Week 56
PD: Change from Baseline in AUC of Acetaminophen to Assess the Delay in Gastric Emptying | Baseline Up to Week 56
PD: Change from Baseline in Time to Peak Drug Concentration (Tmax) of Acetaminophen to Assess the Delay in Gastric Emptying | Baseline Up to Week 56

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - Collaborative Neuroscience Research, LLC, Los Alamitos, California
  - Fortrea Clinical Research Unit, Daytona Beach, Florida
  - Clinical Pharmacology of Miami, Miami, Florida
  - QPS, Springfield, Missouri
  - Fortrea Clinical Research Unit, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3537031 in Overweight, Obese, and Healthy Participants — https://trials.lilly.com/en-US/trial/533078